CLINICAL TRIAL: NCT02464631
Title: To Evaluate the Safety and Efficacy of Sofosbuvir and Ribavirin in Patients With HCV (Genotype 3) Related Decompensated Cirrhosis" - A Randomized Open- Label Study
Brief Title: To Evaluate the Safety and Efficacy of Sofosbuvir and Ribavirin in Patients With HCV (Genotype 3) Related Decompensated Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In view of recent approval of NS5A inhibitors for treatment of hepatitis C such as Declatasvir and Ledipasvir which have proven better efficacy in the HCV cure
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HCV-001
Record Dates: First submitted 2015-05-22; First posted 2015-06-08 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-01

CONDITIONS: HCV Related Cirrhosis
MeSH Terms: interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sofosbuvir + Ribavirin 1 (Active Comparator): Sofosbuvir + Ribavirin x 24 weeks
  Interventions: Drug: Sofosbuvir + Ribavirin 1
- Sofosbuvir + Ribavirin 2 (Experimental): Sofosbuvir + Ribavirin x 36 weeks
  Interventions: Drug: Sofosbuvir + Ribavirin 2
- Sofosbuvir + Ribavirin 3 (Experimental): Sofosbuvir + Ribavirin x 48 weeks
  Interventions: Drug: Sofosbuvir + Ribavirin 3

INTERVENTIONS:
Drug: Sofosbuvir + Ribavirin 1
  Arms: Sofosbuvir + Ribavirin 1
Drug: Sofosbuvir + Ribavirin 2
  Arms: Sofosbuvir + Ribavirin 2
Drug: Sofosbuvir + Ribavirin 3
  Arms: Sofosbuvir + Ribavirin 3

SUMMARY:
In this prospective randomized trial, A Minimum of 300 consecutive patients of decompensated HCV (Hepatitis C Virus) related cirrhosis, presenting to the Institute of Liver and Biliary Sciences hospital will be included and those patients meeting the entry criteria received treatment with 400 mg of Sofosbuvir, administered orally once daily, and Ribavirin administered orally twice daily, with doses determined according to body weight(600 mg daily in patients with a body weight of ≤60 kg,800 mg daily in patients weighing >60 and ≤80 kg, and1000 mg daily in patients with a body weight of >80 kg). Based on the treatment duration, patients would be randomized in either of the 3 treatment groups -

* Group 1 - Sofosbuvir + Ribavirin x 24 weeks
* Group 2 - Sofosbuvir + Ribavirin x 36 weeks
* Group 3 - Sofosbuvir + Ribavirin x 48 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 yrs
* Baseline HCV RNA > 1000 IU/ml
* Cirrhosis with current or prior decompensation
* HCV (Hepatitis C Infection) Genotype 3
* Treatment naïve or treatment experienced

Exclusion Criteria:

* HIV or HBV (Hepatitis B Virus) co-infection
* Recent Variceal bleed
* Pregnancy
* Haemolytic anaemia
* Platelet counts <20,000/ml
* Advanced HCC (Hepatocellular Carcinoma)
* Renal dysfunction, GFR (glomerular filtration rate) < 30 ml/min
* Haemoglobin < 10 g/dl
* MELD (Model for End Stage Liver Disease) >25, CTP (Child-Turcotte-Pugh score) >12
* Post organ transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Primary efficacy end point is SVR 24 defined as HCV RNA <LLOQ (lower limit of quantification) | 48 weeks

SECONDARY OUTCOMES:
The secondary endpoint is any AE (Adverse Event) leading to permanent discontinuation of study drugs. | 3 years
Mortality at 6 months post therapy in all the 3 groups. | 48 weeks
Improvement in the liver function as determined by CTP (Child-Turcotte-Pugh score), MELD (Model for End Stage liver Disease)more than 2 points at 6 months and 1 year. | 48 weeks
Number of new cases of Hepatocellular Carcinoma at end of therapy and at 6 months post therapy in all the 3 groups. | 48 weeks
Reduction in HVPG >20% to baseline after 1 year in all the 3 groups. | 48 weeks
SVR 4 defined as HCV RNA <LLOQ (lower limit of quantification) | 24 weeks
SVR 12 defined as HCV RNA <LLOQ (lower limit of quantification) | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Jindal, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India